CLINICAL TRIAL: NCT03204851
Title: An Open-Label Prospective Pilot Study to Evaluate the Efficacy and Tolerability of Microlyte Ag Pre-Dressing in the Management of Complex Skin Wounds.
Brief Title: Microlyte Dressing in the Management of Wounds
Acronym: Microlyte
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mission Health System, Asheville, NC (Other)
Collaborators: Imbed Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-08-1608
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Wound Heal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Venous Stasis Ulcer (Active Comparator): Venous Stasis Ulcer
  Interventions: Device: Wound Healing
- Pressure Ulcers (Active Comparator): Pressure Ulcers
  Interventions: Device: Wound Healing
- Diabetic Foot Ulcers (Active Comparator): Diabetic Foot Ulcers
  Interventions: Device: Wound Healing
- Wounds from a variety of etiologies (Active Comparator): Wounds from a variety of etiologies
  Interventions: Device: Wound Healing

INTERVENTIONS:
Device: Wound Healing — Microlyte Ag is a class-II medical device cleared by the FDA for prescription and over the counter use in humans with skin wounds.

SUMMARY:
The purpose of this pilot study is to assess the efficacy of Microlyte Ag wound dressing when used in complex skin wounds. Microlyte Ag is a class-II medical device cleared by the FDA for prescription and over the counter use in humans. Primary clinical end point of study is percentage change in wound size from initiation of Microlyte Ag treatment through 90 days or until wound closure. Patient population comprises patients referred to Mission's Wound Healing and Hyperbaric Center for management of their wounds. Targeted enrollment is 100 subjects distributed into 4 study cohorts corresponding to the type of wound treated: venous stasis ulcer (20 patients); diabetic foot ulcer [DFU] (20 patients); pressure ulcer (20 patients); wounds of various other etiologies (40 patients).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age, inclusive
* Venous stasis ulcer, DFU, pressure ulcer, or other wound sufficiently complex as to be referred to Clinical Investigators at Mission's Wound Care and Bariatric Center
* Patient must be competent to consent for self

Exclusion Criteria:

* Patients younger than 18 years of age
* Women who are pregnant or nursing
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10-20 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
percentage change in wound size from initiation of Microlyte Ag treatment through 90 days or until wound closure. | 90 days
  Wound Healing

CONTACTS AND LOCATIONS:
Overall Officials: William Shillinglaw, DO, Study Chair — Mission Health System
Locations (1):
- Mission Health System, Asheville, North Carolina, United States